CLINICAL TRIAL: NCT01975545
Title: Efficacy of the Addition of Silver Nanoparticles to a Fluor Varnish in the Remineralization of Temporary Teeth in Patients With Trisomy 21. Randomized Clinical Trial.
Brief Title: Fluor Varnish With Silver Nanoparticles for Dental Remineralization in Patients With Trisomy 21
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Claudia Butrón Téllez Girón, Claudia Butrón-TéllezGiron, Dent., Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCIC-001
Record Dates: First submitted 2013-09-03; First posted 2013-11-04 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Caries; Dental varnish
MeSH Terms: conditions — Down Syndrome | interventions — Nanoparticles; colloidal silver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluor varnish (Active Comparator): Fluor dental varnish (Fluor Protector, Ivoclar Vivadent, Principality of Liechtenstein)
  Interventions: Drug: Fluor varnish
- Fluor varnish with nanoparticles (Experimental): Fluor dental varnish (Fluor Protector, Ivoclar Vivadent, Principality of Liechtenstein) plus 25% 50 nm silver nanoparticles.
  Interventions: Drug: Fluor varnish with nanoparticles

INTERVENTIONS:
Drug: Fluor varnish — Dental varnish will be applied to one anterior superior teeth in a random side.
  Other Names: Fluor dental varnish
  Arms: Fluor varnish
Drug: Fluor varnish with nanoparticles — Dental varnish with silver nanoparticles will be applied to one anterior superior teeth in a random side.
  Other Names: Fluor dental varnish with silver nanoparticles.
  Arms: Fluor varnish with nanoparticles

SUMMARY:
Patients with trisomy 21 are in greater danger of developing caries. It has been hypothesized that adding silver nanoparticles to fluor varnishes could promote remineralization of the teeth. A split-plot randomized controlled trial will be performed to address this question.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trisomy 21 diagnosed through caryotype
* Age 1 to 6 years old
* Any sex
* White spot present in both upper anterior teeth
* Parental agreement to participate in the study

Exclusion Criteria:

* Hypersensibility to any of the substances used
* Non cooperating patients
* Caries in enamel or dentine in the upper anterior teeth
* Leukemia or diabetes
* Dental fluorosis present

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Remineralization | 3 months
  Remineralization status will be assessed through laser fluorescence of the tooth with a Diagnodent probe (Diagnodent, Kavo, Madrid, Spain)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Pierdant-Pérez, Md, MSc, Study Director — Universidad Autonoma de San Luis Potosí
Locations (1):
- Universidad Autónoma de San Luis Potosí, San Luis Potosí City, San Luis Potosí, Mexico